CLINICAL TRIAL: NCT04027257
Title: Sit Together and Read (STAR) to Improve Reading Skills for Children and Parenting Self-Efficacy for Caregivers: A Pilot Study of Children Affected by Parental Opioid Use and Their Kinship Caregivers
Brief Title: Sit Together and Read (STAR): A Pilot Study of Children and Their Kinship Caregivers
Acronym: STAR-K
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sherine Tambyraja (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor-Investigator, Sherine Tambyraja, Senior Research Specialist, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019B0129
Record Dates: First submitted 2019-06-28; First posted 2019-07-19 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Reading

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to start the intervention immediately after baseline assessment (i.e., treatment) or approximately 15 weeks later after the baseline assessment (i.e., waitlist control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STAR (Experimental): Receive 15-week STAR intervention immediately after pretest.
  Interventions: Behavioral: Sit Together and Read (STAR)
- Waitlist Control (No Intervention): No intervention for the 15 weeks after pretest.

INTERVENTIONS:
Behavioral: Sit Together and Read (STAR) — STAR is an evidence-based home-based shared book reading intervention designed to improve the foundational reading skills of preschoolers who are at risk for reading disabilities.
  Arms: STAR

SUMMARY:
Parental substance use is the second leading cause of foster care placement. As a result, nearly 100,000 Ohio grandparents, family, friends, and neighbors are providing kinship care for children. Kinship caregivers are more likely to be of lower socioeconomic status, report less warmth and respect in their parenting attitudes, and exhibit higher levels of caregiver-child conflict, relative to traditional foster parents. These characteristics, in addition to the trauma associated with exposure to parental drug use, contribute to a significant risk for reading difficulties and lower overall academic achievement for affected children. The objective is to pilot an evidence-based reading intervention in a group of kinship caregivers and children affected by parental opioid use. This work is significant because the investigators aim to improve reading outcomes of children who may otherwise experience substantial difficulty with reading development, and to support kinship caregivers who may otherwise have few resources to promote the reading skills of children placed in their care. The approach will use a randomized (1:1) waitlist controlled trial design to examine the effects of a 15-week kinship caregiver-implemented Sit Together and Read (STAR) intervention for 4-5 year old children being raised by kin as a result of parental opioid use.

DETAILED DESCRIPTION:
Parental substance use is the second leading cause of foster care placement, with nearly 50% of cases involving children under age five years. Fifty percent of all Ohio children taken into child protective services experienced parental drug use, with rates higher than 75% in some Ohio counties. Approximately 100,000 Ohio grandparents and relatives are providing kinship care for children affected by parental drug use.

STAR is an evidence-based home-based shared book reading intervention designed to improve the foundational reading skills of preschoolers who are at risk for reading disabilities. The potential for STAR to positively impact the kinship family is multi-faceted. STAR was developed to accelerate the early reading development of vulnerable children, including those in kinship care. The investigators expect STAR to promote positive caregiver-child interactions and improve kinship caregivers' sense of self-efficacy with respect to supporting the child's reading development. The implementation of the STAR intervention is innovative because it will provide tangible and important financial and material resources that have been effective in improving short- and long-term academic outcomes for children living in low SES environments that may not otherwise be available to kinship families.

The overarching goal is to examine the feasibility and effectiveness of an evidence-based reading intervention in a group of kinship caregivers and children affected by parental opioid use. In this pilot implementation, investigators will enroll up to 50 kinship caregivers and the 4 to 5 year old children in their care to determine the feasibility of the STAR intervention in this population (Aim 1). The investigators will determine the extent to which STAR imparts positive and significant effects on children's foundational reading skills (Aim 2). The investigators will examine the extent to which participation in STAR, and the associated training and supports provided, are associated with positive changes in kinship caregivers' self-efficacy with respect to supporting the reading development of the children in their care (Aim 3). Investigators will meet the objectives of this work by using a randomized (1:1) waitlist controlled trial design. The randomization scheme will be prepared prior to any participant enrollment by a statistician not affiliated with the project. Successful implementation of this work will provide financial and material resources to families in need, while simultaneously engaging kinship families in an evidenced-based intervention that is proven effective at improving young children's reading trajectories.

ELIGIBILITY:
Inclusion Criteria:

* Child 4 years, 0 months to 5 years, 11 months at enrollment
* Child in kinship care
* Child experienced parental opioid use prior to kinship care
* Kinship caregiver willing to attend in-person meetings
* Kinship caregiver willing to read regularly to the child in English for 15 consecutive weeks

Exclusion Criteria:

* NA

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
STAR Log | 15-week intervention period
  Document intensity, defined as occurrence and length of each session and targeted goals within each.
STAR Fidelity Coding Checklist (FCC) | 15-week intervention period
  Document dosage, defined as the volume of explicit targeting of print-related objectives during STAR sessions.
Preschool Word and Print Awareness (PWPA) | 15-week intervention period
  Examines knowledge of 15 print concepts. Scores on this scale range from 0-17, with higher scores indicative of better performance.
Phonological Awareness Literacy Screening-PreK (PALS-PreK) | 15-week intervention period
  Upper and Lower Case Letter Knowledge subtests will identify the number of letters children can name. The range on these subtests is 0-26, with higher scores indicative of better performance. The name writing subtest will assess children's ability to write their own name. The range on this subtest is 0-7, with higher scores indicative of better performance.
Test of Preschool Emergent Literacy (TOPEL) | 15-week intervention period
  The print knowledge subtest will be used to assess children's skills on a variety of print-related tasks, such as distinguishing print from other visual stimuli and identifying alphabet letters. Raw scores on this subtest range from 0-36, with higher scores indicative of better performance
Parenting Sense of Competence Scale | 15-week intervention period
  Assesses kinship caregivers' self-efficacy. Scores on this measure range from 17-102, with higher scores representing a higher parenting sense of competency.

CONTACTS AND LOCATIONS:
Locations (1):
- Email List Servs, Dublin, Ohio, United States

IPD SHARING:
Plan to Share IPD: No